CLINICAL TRIAL: NCT03333525
Title: Does High-Protein High-Fat Meal Increase Postprandial Glucose Concentrations and Meal-Time Insulin Requirements in Patients With Type 1 Diabetes on Basal-Bolus Insulin Regimen: A Randomized Controlled Trial
Brief Title: Does Protein and Fat Content of Meal Increase Glucose Concentrations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Neşe Kaya, Investigator, clinical research, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013/173; KEPAN (Other Grant/Funding Number: Turkish Clinical Enteral Parenteral Nutrition Society); ESPEN Travel Grant (36 th) (Other: The European Society for Clinical Nutrition and Metabolism)
Record Dates: First submitted 2017-10-26; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Fat-protein counting; Type 1 diabetes; Postprandial glucose level
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (4):
- Insulin dose-CARB counting HPM group (Experimental): HPM (high protein meal), contained 36 g protein,17 g fat, 70 g carbohydrate and 11.5 g fiber, was given to the subjects in breakfast meal (08.30 h) in the hospital. The glycaemic index (GI) of meal was 60.40. The insulin dose for meal was calculated according to the carbohydrate counting (insulin-to-carbohydrate ratio-ICR).Capillary blood glucose values were collected and recorded before (0 min) and every 30 minutes thereafter for 240 minutes.
  Interventions: Other: Calculation of insulin dosages for different meals
- Insulin dose-CARB counting HPFM group (Experimental): HPFM (high protein-high fat meal), contained 36 g protein,30 g fat, 70 g carbohydrate and 11.5 g fiber, was given to the subjects in breakfast meal (08.30 h) in the hospital The glycaemic index (GI) of meal was 60.40. The insulin dose for meal was calculated according to the carbohydrate counting (insulin-to-carbohydrate ratio-ICR).Capillary blood glucose values were collected and recorded before (0 min) and every 30 minutes thereafter for 240 minutes.
  Interventions: Other: Calculation of insulin dosages for different meals
- Insulin dose-CARB+FPU counting-HPFM (Experimental): HPFM (high protein-high fat meal), contained 36 g protein,30 g fat, 70 g carbohydrate and 11.5 g fiber, was given to the subjects in breakfast meal (08.30 h) in the hospital. The glycaemic index (GI) of meal was 60.40. The insulin dose for meal was calculated according to the carbohydrate counting plus fat-protein counting (insulin-to-carbohydrate ratio-ICR and fat-protein unit-FPU).Capillary blood glucose values were collected and recorded before (0 min) and every 30 minutes thereafter for 240 minutes.
  Interventions: Other: Calculation of insulin dosages for different meals
- Insulin dose-CARB counting SM group (Active Comparator): SM (standart meal), contained 24 g protein,17 g fat, 70 g carbohydrate and 11.5 g fiber, was given to the subjects in breakfast meal (08.30 h) in the hospital. The glycaemic index (GI) of meal was 60.40. The insulin dose for meal was calculated according to the carbohydrate counting (insulin-to-carbohydrate ratio-ICR and fat-protein unit-FPU).Capillary blood glucose values were collected and recorded before (0 min) and every 30 minutes thereafter for 240 minutes.
  Interventions: Other: Calculation of insulin dosages for different meals

INTERVENTIONS:
Other: Calculation of insulin dosages for different meals — Calculation of insulin dosages For CARB counting meals using insulin-carbohydrate ratio for dosing mealtime boluses. For fat protein counting meal ICR and additionally fat-protein unit were used for dosing of mealtime boluses.

SUMMARY:
The study investigated the effects of fat protein counting (CFP) in addition to carbohydrate (CARB) counting for calculating prandial insulin dosage on blood glucose profile in patients with type 1 diabetes (T1D) on basal-bolus insulin therapy.

DETAILED DESCRIPTION:
In this single center, crossover, randomized, controlled study, control meal (SM: standard meal using carbohydrate counting method) and three test meals (HPM: high protein meal using carbohydrate counting method, HPFM-a: high protein-fat meal using carbohydrate counting method and HPFM-b: high protein-fat meal using carbohydrate and fat-protein counting method) were compared on postprandial early (0-120 minutes), late (120-240 minutes) and total (0-240 minutes) glucose response.

ELIGIBILITY:
Inclusion Criteria:

Subjects:

* had Type1 Diabetes for at least 1 years;
* use multiple dose (basal-bolus) insulin therapy;
* use fast-acting insulin analogs (lispro, glulisine, and aspart) and basal insulin analogs (detemir, glargine);
* daily inslin dose ≥0.5 IU/kg/day.

Exclusion Criteria:

Subjects:

* had any restrictive food intake disorders (eg celiac disease or food allergy);
* had any diabetes complications (eg neuropathy, nephropathy or retinopathy);
* diagnosed for <1 year;
* were using corticosteroid or any medication that could effect gastric emptying;
* did exercise or had hypoglycemia or ketoacidosis within 24 hour before the test meals;
* had overweight or obese (BMI z score: ≥ 1SD and ≥ 2SD respectively);
* had not on follicular or peri-ovulatory phases of their menstrual cycles (for females).

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09-10 (Actual); Primary Completion 2014-02-20 (Actual); Study Completion 2014-02-20 (Actual)

PRIMARY OUTCOMES:
Change Postprandial Glucose Concentrations | 0-240 minutes
  Change from baseline capillary blood glucose values at 240 min after control and test meals consumption.

SECONDARY OUTCOMES:
Postprandial insulin need | [Time Frame: 0-240 minutes]
  Insulin dosage was calculated by FPU (is defined as 100 calories of fat and protein) for HFPM-b meal.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaya N, Kurtoglu S, Gokmen Ozel H. Does meal-time insulin dosing based on fat-protein counting give positive results in postprandial glycaemic profile after a high protein-fat meal in adolescents with type 1 diabetes: a randomised controlled trial. J Hum Nutr Diet. 2020 Jun;33(3):396-403. doi: 10.1111/jhn.12711. Epub 2019 Oct 24. PMID 31647139

DOCUMENTS (1):
  • Study Protocol (2013-05-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT03333525/Prot_000.pdf